CLINICAL TRIAL: NCT02700269
Title: Vanderbilt-Zambia Innovations in Global Health Technologies
Acronym: VZNIGHT
Status: Completed | Type: Observational
Sponsor: Macha Research Trust, Zambia (Other)
Collaborators: Vanderbilt University (Other); National Institutes of Health (NIH) (NIH); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Other Study IDs: MRT15003.2; 5D43TW009348 (NIH); NCT02698774 (obsolete NCT alias)
Record Dates: First submitted 2016-02-25; First posted 2016-03-07 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Malaria Diagnosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Other: mBEADS — Evaluate approaches using magnetic bead capture, isolation, and surface tension valve transfer of biomarkers to improve the sensitivity of already approved malaria RDTs.

SUMMARY:
Investigators will evaluate approaches using magnetic bead capture, isolation, and surface tension valve transfer of biomarkers to process capillary blood in order to improve the sensitivity of already approved Rapid Diagnostic Tests (RDTs) for detection of human malaria infection. Results will be compared to those obtained using unenhanced capillary blood specimens directly applied to approved malaria RDTs. Participants seeking care for possible malaria in Zambia will be recruited to enroll in the study.

ELIGIBILITY:
Inclusion Criteria:

* Individuals giving written informed consent for themselves
* Children under the age of 18 for whom a parent or guardian can give consent
* Individuals seeking care or treatment of suspected or possible malaria
* Individuals being screened as a contact of someone with recent malaria
* Other individuals willing to have their blood tested for malaria

Exclusion Criteria:

* Anyone over 18 unwilling or unable to provide informed consent
* Anyone under 18 who does not have a parent or guardian to give consent
* Anyone between the age of 12 and 18 who does not give assent

Ages: 6 Months to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Those seeking care for suspected malaria in Zambia
Sampling Method: Non-Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Enhancement of malaria RDT to detect low levels of P falciparum parasites | 5 years
  The expected outcome of this research project is to enhance the ability of standard malaria RDTs to detect low levels of Plasmodium falciparum malaria in human capillary blood.

CONTACTS AND LOCATIONS:
Locations (1):
- Macha Research Trust, Choma, Zambia